CLINICAL TRIAL: NCT06363838
Title: Evaluation of Neuromuscular Morphometry of the Vaginal Wall Using Protein Gene Product 9.5 (Pgp 9.5) and Smooth Muscle α-Actin (Sma) in Patients With Posterior Vaginal Wall Prolapse
Brief Title: Evaluation of Neuromuscular Morphometry of the Vaginal Wall
Status: Completed | Type: Observational
Sponsor: Gaziosmanpasa Research and Education Hospital (Other Government)
Collaborators: Ordu University (Other)
Responsible Party: Sponsor
Other Study IDs: ordu eah
Record Dates: First submitted 2024-04-09; First posted 2024-04-12 (Actual); Last update posted 2024-04-12 (Actual); Status verified 2024-03

CONDITIONS: Pelvic Organ Prolapse
Keywords: posterior vaginal wall; prolapse; smooth muscle; actin
MeSH Terms: conditions — Pelvic Organ Prolapse; Prolapse

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- study group: women aged between 40 and 75 years who had not undergone any vaginal surgery and had not undergone any abdominal prolapse surgery were included. Thirty-one women diagnosed with rectocele on examination were included in the study group.Biopsy material was obtained from the epithelium of the posterior wall of the vagina, including the fascia that fits the Ap point. Immunohistochemical staining with Protein Gene Product 9.5 and smooth muscle α-actin was performed in the pathology laboratory. The epithelial thickness measurement and smooth muscle density parameters obtained
- control group: Thirty-one patients who underwent vaginal intervention and hysterectomy for reasons other than rectocele (colposcopy, conization, etc.) without anterior or posterior wall prolapse were included in the control group.Biopsy material was obtained from the epithelium of the posterior wall of the vagina, including the fascia that fits the Ap point. Immunohistochemical staining with Protein Gene Product 9.5 and smooth muscle α-actin was performed in the pathology laboratory. The epithelial thickness measurement and smooth muscle density parameters obtained

SUMMARY:
In this prospective study, women aged between 40 and 75 years who had not undergone any vaginal surgery and had not undergone any abdominal prolapse surgery were included. Thirty-one women diagnosed with rectocele on examination were included in the study group. Thirty-one patients who underwent vaginal intervention and hysterectomy for reasons other than rectocele (colposcopy, conization, etc.) without anterior or posterior wall prolapse were included in the control group.

DETAILED DESCRIPTION:
In this prospective study,who had not undergone any vaginal surgery and had not undergone any abdominal prolapse surgery were included. Thirty-one women diagnosed with rectocele on examination were included in the study group. Thirty-one patients who underwent vaginal intervention and hysterectomy for reasons other than rectocele (colposcopy, conization, etc.) without anterior or posterior wall prolapse were included in the control group. Biopsy material was obtained from the epithelium of the posterior wall of the vagina, including the fascia that fits the Ap point. Immunohistochemical staining with Protein Gene Product 9.5 and smooth muscle α-actin was performed in the pathology laboratory. The epithelial thickness measurement and smooth muscle density parameters obtained with these immunohistochemical stainings were compared between the two groups. The collected data were analyzed using SPSS 23 package program

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 40-75 years
* Patients operated for prolapse
* Patients who did not have prolapse and who would undergo vaginal intervention for other gynecologic reasons were designed to constitute the control group.
* who had not undergone any vaginal surgery, had not undergone any abdominal uterine suspension surgery, had posterior wall prolapse, and for whom surgery was planned.

Exclusion Criteria:

* Patients whose age was not suitable
* who had previously undergone vaginal surgery, who had undergone abdominal surgery and a uterine suspension surgery, who were not suitable for the specified examination conditions
* who had undergone rectocele surgery, urinary incontinence, or bladder surgery

Ages: 40 Years to 75 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — All participants were women because vaginal prolapse was evaluated.
Study Population: The first group included women aged between 40-75 years, who had not undergone any vaginal surgery, had not undergone any abdominal uterine suspension surgery, had posterior wall prolapse, and for whom surgery was planned
Sampling Method: Probability Sample
Enrollment: 62 (Actual)
Dates: Start 2019-12-01 (Actual); Primary Completion 2020-06-25 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
epithelial thickness | one year
  Biopsy material was obtained from the epithelium of the posterior wall of the vagina, including the fascia that fits the Ap point. Immunohistochemical staining with Protein Gene Product 9.5 and smooth muscle α-actin was performed in the pathology laboratory
smooth muscle density | one year
  Biopsy material was obtained from the epithelium of the posterior wall of the vagina, including the fascia that fits the Ap point. Immunohistochemical staining with Protein Gene Product 9.5 and smooth muscle α-actin was performed in the pathology laboratory

CONTACTS AND LOCATIONS:
Overall Officials: HAKAN TİMUR, Study Director — ORDU UNIVERSTY
Locations (1):
- Hakan Timur, Ordu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No